CLINICAL TRIAL: NCT00691431
Title: Comparison of the IntraLaser Femtosecond Laser and Hansatome Mechanical Keratome for Laser In Situ Keratomileusis
Brief Title: IntraLase vs Hansatome Flaps in LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Edward E. Manche, Principal Investigator, Stanford University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-05302008-1190
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2008-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ

INTERVENTIONS:
Device: LASIK

SUMMARY:
This study compared the clinical outcomes between fellow eyes randomized to either IntraLase femtosecond laser-created flaps or Hansatome mechanical keratome-created flaps during wavefront-guided laser in situ keratomileusis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were "T 6.00 D of spherical myopia, "T 3.00 D of refractive astigmatism, stable refraction (less than 0.50D per year of sphere or cylinder), corneal diameter less than 11.0 mm to allow for suction fixation ring, soft contact wearer with discontinuation of wear at least 7 days prior to preoperative evaluation, visual acuity correctable to at least 20/20 in both eyes, more than 21 years of age, ability to participate in follow-up examinations for 12 months after LASIK surgery. In order to fairly compare the visual outcomes of the two keratomes, patients were required to have closely matched eyes, in terms of refractive error. Exclusion Criteria:Exclusion criteria include rigid gas permeable contact lens wearer, severe dry eyes, severe blepharitis, anterior segment pathology (cataracts or corneal scarring or neovascularization within 1 mm of intended ablation zone), recurrent corneal erosion, severe basement membrane disease, progressive or unstable myopia or keratoconus, unstable corneal mires on central keratometry, corneal thickness in which LASIK procedure would result in less than 250 micros or remaining posterior corneal thickness below the flap postoperatively, baseline standard manifest refraction > 0.75 D more minus in sphere power, or a difference of greater than 0.50D in cylinder power compared to baseline standard cycloplegic refraction, two eyes for which the baseline standard cycloplegic refraction differ from each other more than 0.75 in sphere, 0.50 D in cylinder, or have a different type of astigmatism (i.e. with-the-rule) when the cylinder is > 0.50D, or preoperative assessment of ocular topography and/or aberrations indicates that either eye is not suitable candidate for LASIK vision correction procedure (ie forme fruste keratoconus, corneal warpage, or pellucid marginal degeneration), previous intraocular or corneal surgery, and history of herpes zoster or simplex keratitis, patients on systemic corticosteroid or immunosuppressive therapy, immunocompromised subjects or clinically significant atopic disease, connective tissue disease, or diabetes, steroid responder, macular pathology, pregnant or lactating patients, patients with sensitivity to planned study concomitant medications or patients participating in another ophthalmic drug or device clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51
Dates: Start 2004-05; Study Completion 2005-11

PRIMARY OUTCOMES:
Visual acuity

SECONDARY OUTCOMES:
Contrast sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Manche, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States